CLINICAL TRIAL: NCT00118430
Title: Stepped Care for Affective Disorders and Musculoskeletal Pain
Brief Title: Stepped Care for Depression and Musculoskeletal Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH071268 (NIH); R01MH071268 (NIH)
Record Dates: First submitted 2005-07-06; First posted 2005-07-11 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Pain; Depression
Keywords: Back Pain; Knee Pain; Hip Pain; Stepped Care; Antidepressant; Relaxation Techniques; Exercise
MeSH Terms: conditions — Pain; Depression; Back Pain; Motor Activity | interventions — Antidepressive Agents; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stepped Care (Experimental): Stepped care group
  Interventions: Behavioral: Stepped Care; Drug: Antidepressants
- Usual Care (Active Comparator): Treatment as usual group
  Interventions: Drug: Usual Care
- No Treatment (No Intervention): Participants without depression group

INTERVENTIONS:
Behavioral: Stepped Care — Stepped care will consist of 12 weeks of antidepressant therapy, followed by a pain self-management program (PSMP) in those who fail to achieve both a good pain and global clinical response to antidepressant therapy. Treatment will be delivered by a nurse depression-pain clinical specialist (DPCS) who will be trained in providing both components of the stepped care treatment. The DPCS will meet weekly to review cases with a physician-investigator who will also be available to discuss any management issues that arise between the weekly case meetings. All participants will have six clinical contacts with the DPCS during the acute treatment phase and two clinical contacts during the continuation phase to assess medication adherence, adverse effects, and depression response.
  Arms: Stepped Care
Drug: Antidepressants — Participants will be assigned to one of the following antidepressant regimens: venlafaxine (37.5 mg, increased to 75, 150, 225 mg); duloxetine (60 mg, increased to 120 mg); fluoxetine (20 mg, increased to 30 to 40 mg); sertraline (50 mg, increased to 100 to 150 mg); citalopram (20 mg, increased to 30 to 40 mg); paroxetine (20 mg, increased to 30 to 40 mg); or nortriptyline (25 mg, increased to 50 to 75 mg).
  Arms: Stepped Care
Drug: Usual Care — This group will receive care as usual from their providers and completes the same outcome assessments as the stepped care group.
  Other Names: Standard Care
  Arms: Usual Care

SUMMARY:
This study will evaluate the effectiveness of a stepped care approach in treating depression and reducing pain.

DETAILED DESCRIPTION:
In the United States, pain accounts for nearly 20% of all primary health care visits. In the majority of cases, the pain is musculoskeletal and primarily affects the lower back, hips, and knees. Studies have shown that at least one-third of patients with pain also suffer from depression. It has not been determined whether treatments for depression are effective in patients with comorbid pain and depression. The "Stepped Care for Affective Disorders and Musculoskeletal Pain" (SCAMP) study will determine the most effective treatment for patients with pain and depression.

This study will last 12 months and will comprise depressed and nondepressed participants. Nondepressed participants will receive no treatment. Depressed patients will be randomly assigned to receive standard of care or stepped care for 12 weeks. Standard of care may include cognitive therapy, antidepressant treatment, or other treatments. The stepped care group will receive 12 weeks of antidepressant treatment. Participants who respond to antidepressant treatment will continue their treatment for the duration of the study. Participants who do not respond to the treatment after 12 weeks will receive 6 weekly pain self-management sessions. During these sessions, an educator will teach participants how to manage their pain through exercise and relaxation techniques. Self-report scales and questionnaires will be used to assess participants' pain, depressive symptoms, health care usage and costs, and quality of life. Depressed participants will undergo assessments at study start and at Months 1, 3, 6, and 12. Nondepressed participants will undergo assessments at study start and at Months 3 and 12.

Study hypotheses: 1) Stepped care is more effective than usual care in improving depression and pain. 2) Stepped care is more effective than usual care in improving health-related quality of life, negative pain beliefs and behaviors, reduced opiate use, and health care costs. 3) Patients with musculoskeletal pain who are not depressed at baseline will have an incidence of depression less than 20% over 12 months of follow-up, characteristics that can be identified as risk factors for incident depression, baseline characteristics distinguishing them from depressed patients, and better pain and health status outcomes, compared to depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe pain in the back, hips, or knees for at least 3 months prior to study entry
* History of or current use of at least one medication for pain
* English-speaking

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Schizophrenia or other psychotic disorders
* Receiving disability benefits for pain
* Anticipated life expectancy less than 12 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-09; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Kroenke, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Medical Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data has been published in multiple publications. Should others wish access to data for publication reasons, we are willing to share

REFERENCES:
- [Derived] Dube P, Kurt K, Bair MJ, Theobald D, Williams LS. The p4 screener: evaluation of a brief measure for assessing potential suicide risk in 2 randomized effectiveness trials of primary care and oncology patients. Prim Care Companion J Clin Psychiatry. 2010;12(6):PCC.10m00978. doi: 10.4088/PCC.10m00978blu. PMID 21494337
- [Derived] Kroenke K, Bair MJ, Damush TM, Wu J, Hoke S, Sutherland J, Tu W. Optimized antidepressant therapy and pain self-management in primary care patients with depression and musculoskeletal pain: a randomized controlled trial. JAMA. 2009 May 27;301(20):2099-110. doi: 10.1001/jama.2009.723. PMID 19470987

RESULTS

PARTICIPANT FLOW:
Groups:
- Stepped Care: Stepped care group
  Stepped Care: Stepped care will consist of 12 weeks of antidepressant therapy, followed by a pain self-management program (PSMP) in those who fail to achieve both a good pain and global clinical response to antidepressant therapy. Treatment will be delivered by a nurse depression-pain clinical specialist (DPCS) who will be trained in providing both components of the stepped care treatment. The DPCS will meet weekly with a physician-investigator to review cases, the physician-investigator will be available at all times to discuss any management issues that arise between the weekly case meetings. All participants will have six clinical contacts with the DPCS during the acute treatment phase and two clinical contacts during the continuation phase to assess medication adherence, adverse effects, and depression response
  Antidepressants: Participants will be assigned to one of the following antidepressant regimens: venlafaxine (37.5 mg, increased to 75, 150, 225 mg
Period: Overall Study
Arm/Group | Stepped Care | Usual Care | No Treatment
Started | 123 | 127 | 250
Completed | 102 (123 included in primary analysis due to repeated measures and interim 1,3 and 6 month assessments) | 103 (127 included in primary analysis due to repeated measures and interim 1,3 and 6 month assessments) | 222
Not Completed | 21 | 24 | 28
Not completed — Withdrawal by Subject | 6 | 2 | 0
Not completed — Lost to Follow-up | 15 | 22 | 28

BASELINE CHARACTERISTICS:
Groups:
- Stepped Care: Stepped care group
  Stepped Care: Stepped care will consist of 12 weeks of antidepressant therapy, followed by a pain self-management program (PSMP) in those who fail to achieve both a good pain and global clinical response to antidepressant therapy. Treatment will be delivered by a nurse depression-pain clinical specialist (DPCS) who will be trained in providing both components of the stepped care treatment. The DPCS will meet weekly to review cases with a physician-investigator who will also be available to discuss any management issues that arise between the weekly case meetings. All participants will have six clinical contacts with the DPCS during the acute treatment phase and two clinical contacts during the continuation phase to assess medication adherence, adverse effects, and depression response.
  Antidepressants: Participants will be assigned to optimization of venlafaxine, duloxetine, fluoxetine, sertraline, citalopram, paroxetine, or nortriptyline.
- Total: Total of all reporting groups
Arm/Group | Stepped Care | Usual Care | No Treatment | Total
Number analyzed (Participants) | 123 | 127 | 250 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (12.6) | 55.8 (11.1) | 62.5 (14.1) | 59.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 63 | 127 | 259
  Male | 54 | 64 | 123 | 241
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 42 | 49 | 100 | 191
  White | 75 | 76 | 140 | 291
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 123 | 127 | 250 | 500
HSCL-20 depression severity [Mean (Standard Deviation); unit: units on a scale] — This scale consists of 20 items, each scored from 0 (lowest) to 4 (highest or worst). The scale score is the average of the 20 items. Therefore, the HSCL-20 depression severity score can range from 0 (no depression) to 4 (highest or worst depression)
  units on a scale | 1.8 (0.7) | 1.9 (0.6) | 0.7 (0.5) | 1.3 (0.8)
Brief Pain Inventory severity [Mean (Standard Deviation); unit: units on a scale] — The BPI severity scale is a 4-item scale with each item scored from 0 (no pain) to 10 (worst pain imaginable). The scale score is the average of the 4 items and thus can range from 0 (no pain) to 10 (worst or more severe pain)
  units on a scale | 6.2 (1.8) | 6.1 (1.8) | 5.4 (1.8) | 5.8 (1.8)
Brief Pain Inventory interference [Mean (Standard Deviation); unit: units on a scale] — The BPI interference scale consists of 7 items, each scored from 0 (no interference) to 10 (complete interference), and the total score is the average of the 7 individual item scores. Therefore, the BPI interference score can range from 0 (lowest pain) to 10 (worst or highest pain).
  units on a scale | 6.8 (2.2) | 7.1 (2.0) | 4.8 (2.2) | 5.9 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory Interference
Description: The BPI interference scale consists of 7 items, each scored from 0 (no interference) to 10 (complete interference), and the total score is the average of the 7 individual item scores. Therefore, the BPI interference score can range from 0 (lowest pain) to 10 (worst or highest pain).
Time Frame: Measured at Year 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care | Usual Care | No Treatment
Number analyzed (Participants) | 123 | 127 | 250
units on a scale | 5.0 (2.8) | 6.5 (2.4) | 4.6 (2.4)
Statistical Analysis 1: Comparison: Stepped Care vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This reported p-value was calculated (and does not merely represent the threshold for significance

2. Primary Outcome: HSCL-20 Depression Severity
Description: This scale consists of 20 items, each scored from 0 (lowest) to 4 (highest or worst). The scale score is the average of the 20 items. Therefore, the HSCL-20 depression severity score can range from 0 (no depression) to 4 (highest or worst depression)
Time Frame: Measured at Year 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care | Usual Care | No Treatment
Number analyzed (Participants) | 123 | 127 | 250
units on a scale | 1.1 (0.7) | 1.7 (0.7) | 0.8 (0.6)
Statistical Analysis 1: Comparison: Stepped Care vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — This reported p-value was calculated (and does not merely represent the threshold for significance

3. Secondary Outcome: Graded Chronic Pain Scale Disability Score
Description: This scale ranges from 0 (no pain-specific disability) to 100 (highest or worst pain-specific disability)
Time Frame: Measured at Year 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care | Usual Care | No Treatment
Number analyzed (Participants) | 123 | 127 | 250
units on a scale | 52.5 (31.6) | 66.1 (27.3) | 44.8 (29.6)
Statistical Analysis 1: Comparison: Stepped Care vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

4. Secondary Outcome: Primary Care Visits
Time Frame: Measured at Year 1
Population: The no treatment group did not have depression and was followed simply as a cohort and not part of the clinical trial. Therefore we did not measure this secondary outcome of primary care visits in the no treatment group.
Measure: Mean (Standard Deviation); unit: number of primary care visits
Arm/Group | Stepped Care | Usual Care
Number analyzed (Participants) | 123 | 127
number of primary care visits | 6.3 (5.8) | 5.9 (5.3)
Statistical Analysis 1: Comparison: Stepped Care vs Usual Care; Test type: Superiority or Other; p < 0.001, Poisson

ADVERSE EVENTS:
Description: The no treatment group did not have depression and was simply followed as a cohort and were not part of the actual clinical trial. Thus, adverse events were not assessed in this group.
Arm/Group | Stepped Care | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/127
Other Adverse Events (participants affected / at risk) | 0/123 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No